CLINICAL TRIAL: NCT02785822
Title: Randomized, Single Blind, Prospective Clinical Study to Compare hFSH-HP (Fostipur) and hMG-HP(Meriofert) in Patients With Polycystic Ovary Under a IVF/ICSI Cycle.
Brief Title: Study to Compare hFSH-HP (Fostipur) and hMG-HP(Meriofert) in Patients With Polycystic Ovary Under a IVF/ICSI Cycle.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Programa de Reproducción Asistida F. Puigvert - HSCSP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-FOS-2016-01
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Reproductive Techniques, Assisted
MeSH Terms: conditions — Polycystic Ovary Syndrome; Helping Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fostipur (Active Comparator)
  Interventions: Drug: hFSH-HP
- Meriofert (Experimental)
  Interventions: Drug: hMG-HP

INTERVENTIONS:
Drug: hMG-HP — Ovarian stimulation with hMG-HP (150 IU / day)
  Other Names: Meriofert
  Arms: Meriofert
Drug: hFSH-HP — Ovarian stimulation with hFSH-HP (150 IU / day)
  Other Names: Fostipur
  Arms: Fostipur

SUMMARY:
Polycystic ovary occurs in 15-20% of the population will be submitted to TRA. Whether it is associated with other signs or symptoms (polycystic ovarian syndrome) as if presented in isolation, its therapeutic management has special connotations sometimes favoring the low response although the standard is the tendency to hyperresponsiveness.

Although there are studies comparing the combination of FSH and LH and FSH in controlled hyperstimulation of these patients, there are no previous prospective randomized studies comparing administration of urinary FSH (hFSH-HP) with a combination of FSH and HCG (HMG HP).

Therefore the aim of this study is to prove that both drugs are comparable in the treatment of these patients. The test substances are marketed in Spain (Fostipur and Meriofert, respectively) with an indication for use in these patients. In this study both medicines will be administered in a randomized way under the usual conditions in which it is used in routine clinical practice to compare the quantity of mature oocytes respect to the total oocytes obtained, as a primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 18 and 38 years (inclusive)
* Women with a BMI under 30 kg / m2
* Diagnosis of polycystic ovary syndrome (according to criteria of Rotterdam)
* Women who want pregnancy
* Basal basal FSH levels under or equal 10 IU / l
* Infertility justify treatment with in vitro fertilization / intracytoplasmic sperm injection
* To be included in a protocol with GnRH antagonist
* Presence of both ovaries and uterus able to support embryo implantation and pregnancy
* Absence of pregnancy before starting ovarian stimulation
* Written consent

Exclusion Criteria:

* Severe male factor not allowing an in vitro fertilization / intracytoplasmic sperm injection with ejaculated sample
* Patients with low ovarian reserve
* Important endocrine-metabolic systemic diseases affecting pituitary, thyroid, adrenals, pancreas, liver or kidney
* HIV seropositivity
* To have frozen embryos from previous cycles of assisted reproduction
* Undiagnosed vaginal haemorrhage
* Poor response in previous cycles of in vitro fertilization with standard stimulation protocols
* Pregnancy, lactation or contraindication to get pregnant
* Malformations of the sexual organs incompatible with pregnancy
* History of allergy to gonadotrophin preparations or its excipients
* Alcohol, drugs or psychotropic addiction
* Concurrent participation in another study
* Previous history of severe hyperstimulation syndrome
* Concomitant medication that may interfere with the study medication: different hormonal treatments used in the study, other thyroid hormones, antipsychotics, anxiolytics, hypnotics, sedatives, chronic treatment with inhibitors of prostaglandin

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Quantity of mature oocytes respect to the total oocytes | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Espinos, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Fundació Puigvert, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona